CLINICAL TRIAL: NCT01112046
Title: Endoscopic Submucosal Dissection Versus Laparoscopic Resection for Early Colorectal Neoplasms: A Prospective Randomized Trial
Brief Title: Endoscopic Submucosal Dissection Versus Laparoscopic Resection for Early Colorectal Neoplasms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: United Christian Hospital (Other); Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2009.625
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Colorectal Neoplasms
Keywords: Early colorectal neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic submucosal dissection (Experimental)
  Interventions: Procedure: Endoscopic submucosal dissection
- Laparoscopic resection (Active Comparator)
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — Endoscopic treatment (performed under conscious sedation) using specific endoscopic knives
  Other Names: ESD
  Arms: Endoscopic submucosal dissection
Procedure: Laparoscopic resection — Surgical treatment performed under general anesthesia
  Arms: Laparoscopic resection

SUMMARY:
This is a prospective randomized trial that aimed to compare the short-term clinical outcomes and systemic inflammatory/cytokine responses of endoscopic submucosal dissection versus laparoscopic resection for early colorectal neoplasms that are not amenable to en bloc endoscopic resection with conventional techniques.

DETAILED DESCRIPTION:
Colonoscopy plays an increasingly important role in the diagnosis and treatment of colorectal pathologies. The recent progress in endoscopic technologies and interest in colorectal cancer screening have enabled the diagnosis of a larger number of early colorectal neoplasms, including benign polyps and early cancers. Colonoscopic polypectomy remains the cornerstone of therapy for the majority of colorectal polyps and helps prevent colorectal cancer. However, if colorectal neoplasms are too large or cannot be removed "en bloc" endoscopically, operative procedures are required to reduce risks of incomplete removal and local recurrence. Laparoscopic resection represents a minimally invasive alternative for treating colorectal neoplasms that are not amenable to en bloc endoscopic resection. However, laparoscopic surgery has to be done under general anesthesia, is associated with operative morbidity, and is expensive.

Endoscopic submucosal dissection (ESD) is a revolutionary endoscopic procedure that enables en bloc resection of large gastrointestinal tumors, irrespective of the size of the lesion. ESD, which was pioneered in Japan for the treatment of early gastric neoplasms, has now been successfully applied to the colon and rectum. ESD has been shown by recent studies to be a safe and effective resection technique for large early colorectal neoplasms. However, no report can be found in the literature comparing ESD and laparoscopic resection for early colorectal neoplasms that are not amenable to en bloc endoscopic resection with conventional techniques. Furthermore, it remains unclear whether ESD is less invasive than laparoscopic surgery in terms of systemic inflammatory and cytokine responses, and all these may have implications for cancer recurrence.

We propose to conduct a prospective randomized trial to compare the short-term clinical outcomes and systemic inflammatory/cytokine responses of ESD versus laparoscopic resection for early colorectal neoplasms that are not amenable to en bloc endoscopic resection with conventional techniques. The overall costs of the two therapeutic approaches will also be compared. Findings of this proposed project may provide evidence-based clarification of the efficacy and safety of ESD in treating early colorectal neoplasms. We hypothesize that ESD is associated with lower morbidity, earlier recovery, shorter hospital stay, and lower costs when compared with laparoscopic resection. A faster recovery and earlier discharge after ESD may reduce financial burden to the hospital and health care system. The results of this proposed project may have a significant impact on the future treatment strategy for early colorectal neoplasms, and may provide new insights into the systemic inflammatory responses of ESD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with early colorectal neoplasms >/= 2 cm in size in the colon or upper rectum (>/= 15 cm above the anal verge) that are deemed not feasible for en bloc resection with conventional polypectomy or EMR as judged by 2 experienced endoscopists,
* Age of patients >18 years,
* Patients with American Society of Anesthesiologists (ASA) grading I-III,
* Informed consent available

Exclusion Criteria:

* Presence of endoscopic signs of massive submucosal invasion (including excavated/depressed morphology or Kudo's pit pattern Type V),
* Endosonographic evidence of deep invasion,
* Unfavorable histopathologic features on biopsy (including mucinous cancer, poor differentiation, and gross submucosal invasion),
* Patients with other synchronous colorectal neoplasms in addition to the index neoplasm that are not amenable to complete endoscopic removal, neoplasms occupying more than half circumference of the colonic wall,
* Patients with recurrence from previous endoscopic mucosal resection or ESD,
* Patients with known metastatic disease,
* Patients with previous history of abdominal surgery, and patients with non-correctable coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2010-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Short-term morbidity | Up to 1 month

SECONDARY OUTCOMES:
Systemic cytokine and C-reactive protein levels | Up to 5 days
  Measured at 2 hours, 8 hours, 24 hours, 48 hours, and 5 days after ESD/surgery
Post-ESD/surgery recovery | Up to 1 month
  Time to resume normal diet, time to walk independently, and duration of hospital stay
Quality of life | Up to 1 year
  Measured by Short Form-36 (SF-36) and European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaires at 3, 6, 9, and 12 months after ESD/surgery
Direct and indirect medical costs | Up to 1 year
Local recurrence | Within 5 years after ESD/surgery

CONTACTS AND LOCATIONS:
Overall Officials: Simon SM Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China